CLINICAL TRIAL: NCT00176943
Title: Phenotype and Cytokine Production Characteristics of T Cells From Alopecia Areata Scalp Skin Before and After Aldara 5% Cream Using Flow Cytometry
Brief Title: Characteristics of T Cells From Alopecia Areata Scalp Skin Before and After Treatment With Aldara 5%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hordinsky, Maria K., MD (Individual)
Collaborators: National Alopecia Areata Foundation (Other)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0009M64941
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aldara Cream 5%

SUMMARY:
It is thought that alopecia areata occurs as the result of an inappropriate response of the body's own immune system to certain substances in or around the hair follicle. We will be examining the efficacy of Aldara Cream 5% in treating extensive alopecia areata and observe its affect on the hair follicle.

DETAILED DESCRIPTION:
We will examine how the application of Aldara Cream 5% daily for 6 months will affect the hair follicle and the inflammation present in the skin of patients with alopecia areata. In the study we will obtain additional scalp biopsies to examine how the drug affects the quality and state of activity of the immune cells in the biopsy specimens. This type of information will provide data about the behavior of these inflammatory cells in mediating the hair loss associated with alopecia areata and how this behavior may be effected by Aldara Cream 5% treatment. Such information may be valuable to the successful management of alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health.
* No topical or systemic treatment for alopecia areata for at least 2 weeks prior to study initiation.
* Must be at least 18 years of age and older
* Will have to have extensive scalp alopecia areata (>95% involvement) of less than 2 years duration.
* Willing to refrain from other alopecia areata treatments during the course of the study.
* Will have to agree to shampoo their scalp daily with Free and Clear shampoo. Participant in "Aldara for the Treatment of Extensive Alopecia Areata" study.

Exclusion Criteria:

* History of any illness or condition that in the opinion of the investigator might confound the results of the study or pose additional risk to the patient
* Significant abnormalities on screening clinical evaluation.
* Previous use of Aldara Cream 5%.
* A history of drug or alcohol abuse.
* Use of UV radiation including tanning beds and PUVA therapy for treatment of acne, psoriasis, or any other skin condition within 2 months prior to study initiation.
* Use of systemic or topical glucocorticoids, corticosteroids, estrogenic, progestogenic, androgenic or antiandrogen drugs, cyclosporine, FK506 or immunotherapy with DNCB,SADBE or DCP within 6 months of study initiation.
* Alterations in thyroid medication within 6 weeks of study initiation. Pregnant or nursing females. Not participating in the "Aldara for the Treatment of Extensive Alopecia Areata" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2000-10; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
To determine the phenotypic characteristics of T lymphocytes infiltrating scalp dermis and epidermis in patients with extensive alopecia areata before and after treatment with Aldara Cream 5% an immunomodulatory agent.

SECONDARY OUTCOMES:
To further characterize the functional potential of these cells using the nascent technology of intracellular cytokine staining.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Marna Ericson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States